CLINICAL TRIAL: NCT06060821
Title: Construct Validity and Reliability of the 2-minute Step Test in Patients With Lumbar Spinal Stenosis
Brief Title: Validity and Reliability of the 2-minute Step Test in Patients With Lumbar Spinal Stenosis
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstPRMTRH1
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Spinal Stenosis
Keywords: Exercise test; Spinal stenosis; Physical fitness
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study was to investigate the validity and reliability of the 2 Minute Step Test (2MST) in patients with symptomatic degenerative lumbar spinal stenosis and to explore its correlation with objective assessment methods, namely the 2 Minute Walk Test (2MWT) and the 6 Minute Walk Test (6MWT).

DETAILED DESCRIPTION:
This cross-sectional study will include 55 volunteers aged 18-80 years who present to the Istanbul Physical Medicine and Rehabilitation Training and Research Hospital outpatient clinics and are diagnosed with Lumbar Spinal Stenosis (LSS) through MRI. The demographic characteristics of the patients will be recorded, and their walking distances will be inquired about. The severity of the disease will be determined by examining the levels of stenosis on lumbar MRI scans. All patients will be initially assessed using the 2MST (2-Minute Step Test), 2MWT (2-Minute Walk Test), 6MWT (6-Minute Walk Test), VAS (Visual Analogue Scale), and ODI (Oswestry Disability Index). To measure test-retest reliability, the 2MST will be administered again with a 7-day interval between assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 who have been diagnosed with lumbar spinal stenosis based on magnetic resonance images.

Exclusion Criteria:

* Uncontrolled hypertension
* Decompensated heart failure
* Presence of systemic diseases affecting lower extremity functions
* Presence of degenerative diseases affecting lower extremity functions
* Peripheral artery disease causing vascular claudication
* Psychiatric illness
* Neuromuscular disease
* Pregnancy
* Cognitive impairment

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-80 who have been diagnosed with lumbar spinal stenosis based on magnetic resonance images.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
2-minute step test | Baseline and Day 7
  The patient was instructed to lift their knees to the minimum marked level and take as many steps as possible in place for a duration of two minutes.

SECONDARY OUTCOMES:
6-minute walk test | Baseline and Day 7
  The distance the patient walked for six minutes was measured.
2-minute walk test | Baseline and Day 7
  The distance the patient walked for two minutes was measured.
Oswestry Disability Index | Baseline and Day 7
  This is a patient-reported outcome measure used by clinicians and researchers to quantify disability related to low back pain: Higher scores indicate worse functional status.
Visual Analogue Scale | Baseline and Day 7
  Pain score; higher scores indicate higher pain levels.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Kesiktas, MD, Study Chair — İstanbul Physical Therapy Rehabilitation Training & Research Hosptial
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paker N, Sirin Ahisha B, Kesiktas N, Bugdayci ND, Soluk Ozdemir Y. Construct validity and reliability of the 2-minute step test in patients with lumbar spinal stenosis. Disabil Rehabil. 2025 Jul;47(14):3708-3713. doi: 10.1080/09638288.2024.2428824. Epub 2024 Nov 19. PMID 39563102